CLINICAL TRIAL: NCT05217797
Title: The GLasses Against Transmission of SARS-CoV-2 (COVID-19) in the communitY (GLASSY) Trial: A Pragmatic Randomized Trial
Brief Title: Glasses Against Transmission of SARS-CoV-2 (COVID-19) in the Community
Acronym: GLASSY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Institute of Public Health (Other Government)
Collaborators: University of Basel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P360-22/00592
Record Dates: First submitted 2022-01-31; First posted 2022-02-01 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: COVID-19; Respiratory Tract Infections
Keywords: COVID-19 Prevention Protection
MeSH Terms: conditions — COVID-19; Respiratory Tract Infections

STUDY DESIGN:
Intervention Model Description: Sequence generation We will use a simple 1:1 randomization by means of computer-generated random numbers.
  The allocation will be concealed as the participant themselves will be directly informed of their allocation as soon as they have agreed to take part in the trial and have completed the online consent form. Generation of allocation sequence, enrolment of participants and assignment of participants will all be handled by the digital recruitment platform.
Masking Description: No blinding was feasible, except for in the analysis phase. One member of our team (A.H.) provided the chief analyst (I.H.E.) with a data file in which group allocation was blinded. The chief analyst presented the main results to the project team members, who were also blinded to the group allocation (and data on use of glasses). We discussed how we would interpret the findings depending on whether one group or the other was the intervention group, and we prepared a short report that we posted online before unblinding ourselves to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glasses (Experimental): Participants in the experimental arm are asked to wear glasses (sunglasses or other glasses) when outside their home and close to others (e.g. on public transport, in shopping centres etc.).
  Interventions: Behavioral: Wearing glasses (any type)
- Not glasses (No Intervention): Participants in no interventions arm are asked to not wear glasses (sunglasses or other glasses) when outside their home and close to others (e.g. on public transport, in shopping centres etc.).

INTERVENTIONS:
Behavioral: Wearing glasses (any type) — Participants are asked to wear glasses in public spaces.
  Arms: Glasses

SUMMARY:
In this trial the researchers plan to recruit 25,000 volunteers to be randomly allocated either wearing sunglasses or ordinary glasses in public spaces where they are close to other people, or not wear glasses in such circumstances. For each participant the trial period is 2 weeks, after which they will be asked to complete a brief questionnaire which includes questions about results of COVID-19 tests during the trial period.

DETAILED DESCRIPTION:
A systematic review of observational studies indicated that eye protection may be an effective measure to prevent SARS-CoV-2 infections. Randomized trials are needed to assess whether the observed associations are caused by protection of the eye or confounding factors such as other systematic differences between users and non-users of eye protection, co-interventions, or changes in COVID-19 incidence when comparisons were done over time.

This is a pragmatic, virtual, parallel group, 1:1 randomized, superiority trial. The researchers will recruit and randomize participants via an online portal. The trial will be fully remote and virtual without any personal interaction between investigators and participants. All members of the public are eligible who confirm that they are at least 18 years of age, do not regularly wear glasses, have not contracted COVID-19 since December 15th 2021, and are willing to be randomized to wear, or not wear glasses in public when close to other people, for a 2-week period. Persons who are dependent on visual aids but typically use contact lenses are eligible. The participants will be randomized (1:1) to wear glasses (sunglasses or other types of glasses) in public spaces when close to others (public transport, shopping centers etc.), or to the control group. The control group will be asked not to wear glasses in public spaces when close to others. The primary outcome is positive test for COVID-19.

The researchers aim to include about 25,000 participants to have a statistical power of 80% to detect a relative risk reduction of 25% for the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* owns or can borrow glasses that can be used (e.g. sun-glasses)
* willing to be randomized to wear, or not wear glasses outside the home when close to others, for a 2-week period.
* provides informed consent

Exclusion Criteria:

* does regularly wear glasses (contact lenses are accepted)
* contracted COVID-19 after December 15th 2021.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3717 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Positive test for SARS-CoV-2 | Days 3 to 17 after start of trial period.
  The investigators will compare the incidence of notified cases of COVID-19 (i.e. registered positive SARS-CoV-2 tests).

SECONDARY OUTCOMES:
Health care use for respiratory symptoms | Day 1 to 28
  Routinely collected data (Norwegian Registry for Primary Health Care (KPR) and Norwegian Patient Registry (NPR) databases)
Health care use for injuries health care use (all causes) from day 1 to day 21 (data source: KPR and NPR | Day 1 to 21
  Routinely collected data (KPR and NPR databases)
Health care use (all causes) | Day 1 to 21
  Routinely collected data (KPR and NPR databases)
Any positive COVID-19 test result | Day 1 to 17
  Self report
Respiratory symptoms | Day 1 to 17
  Self report
Health care use for respiratory symptoms | Day 1 to 17
  Self report
Health care use for injuries | Day 1 to 17
  Self report
Health care use (all causes) | Day 1 to 17
  Self report

CONTACTS AND LOCATIONS:
Overall Officials: Atle Fretheim, PhD, Principal Investigator — Head of Centre for Epidemic Interventions Research (CEIR)
Locations (1):
- Norwegian Institute of Public Health, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
From protocol:
  The researchers intend to give full access to the full protocol, participant-level dataset, and statistical code, to anyone who is interested, after securing that the dataset is fully anonymized.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: The investigators expect to be able to share unidentifiable dataset with partners inside the European Union (EU) by May 2022, and an anonymous dataset for wide distribution at a later stage.
Access Criteria: Data that are not fully anonymized will only be shared within the EU (due to data protection regulations).

REFERENCES:
- [Result] Fretheim A, Elgersma IH, Helleve A, Elstrom P, Kacelnik O, Hemkens LG. Effect of Wearing Glasses on Risk of Infection With SARS-CoV-2 in the Community: A Randomized Clinical Trial. JAMA Netw Open. 2022 Dec 1;5(12):e2244495. doi: 10.1001/jamanetworkopen.2022.44495. PMID 36454571